CLINICAL TRIAL: NCT03127839
Title: The Effectiveness of Exercise and Education Type in Patients With SubAcromial Pain Syndrome (SAPS): A Randomized Controlled Trial
Brief Title: Type of Exercise and Education in Patients With SubAcromial Pain Syndrome
Acronym: SAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director of Clinical Outcomes Research at the Center for the Intrepid, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2017.018d
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Shoulder Pain
Keywords: Exercise; Pain Neuroscience Education; Physical Therapy; Subacromial Pain; Rotator Cuff
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eccentric Strengthening Exercise (Active Comparator): Patients will be asked to complete at least 6 outpatient PT sessions over a 4-week period. This will include an individualized impairment-focused approach, utilizing eccentric strengthening exercises of the rotator cuff to address any impairments or reinforce any standard of care manual treatment. Patients will also be given a home exercise program with instructions so that they can perform the eccentric strengthening exercises daily at home.
  Interventions: Procedure: Eccentric Strengthening
- Traditional Strengthening Exercise (Active Comparator): Patients will be asked to complete at least 6 outpatient PT sessions over a 4-week period. This will include an individualized impairment-focused approach, utilizing traditional rotator cuff strengthening exercises to address any impairments or reinforce any standard of care manual treatment. Patients will also be given a home exercise program with instructions so that they can perform the traditional rotator cuff strengthening exercises daily at home.
  Interventions: Procedure: Traditional Strengthening
- Eccentric Exercise + pain education (Active Comparator): In addition to the treatment provided in the "Eccentric Exercise" Arm patients will receive additional self-management training education focused on neuroscience of pain principles.
  This will include e a 5-minute video called "Understanding pain in less than 5 minutes, and what to do about it!", or aka "explain pain" video. The patients will also receive an interactive education booklet and review session with their PT, a series of weekly e-mails that reinforce key components of the booklet and video; and reinforcing messages when in the clinic doing their exercises.
  Interventions: Procedure: Eccentric Strengthening; Behavioral: Pain education
- Traditional Exercise + pain education (Active Comparator): In addition to the treatment provided in the "Traditional Exercise" Arm patients will receive additional self-management training education focused on neuroscience of pain principles.
  This will include e a 5-minute video called "Understanding pain in less than 5 minutes, and what to do about it!", or aka "explain pain" video. The patients will also receive an interactive education booklet and review session with their PT, a series of weekly e-mails that reinforce key components of the booklet and video; and reinforcing messages when in the clinic doing their exercises.
  Interventions: Procedure: Traditional Strengthening; Behavioral: Pain education

INTERVENTIONS:
Procedure: Eccentric Strengthening — Use of eccentric strengthening exercises in treatment plan during visits and at home.
  Arms: Eccentric Exercise + pain education; Eccentric Strengthening Exercise
Procedure: Traditional Strengthening — Use of traditional strengthening exercises in treatment plan during visits and at home.
  Arms: Traditional Exercise + pain education; Traditional Strengthening Exercise
Behavioral: Pain education — Addition of pain neuroscience-focused education in addition to strengthening exercise program
  Other Names: Pain Neuroscience Education; Therapeutic Neuroscience Education
  Arms: Eccentric Exercise + pain education; Traditional Exercise + pain education

SUMMARY:
Patients seeking care for shoulder pain will be recruited to enroll will be randomized to one of four combined treatment groups; eccentric or traditional strengthening alone and eccentric or traditional strengthening with pain neuroscience education. Patients will be followed for 1 year.

DETAILED DESCRIPTION:
Patients seeking care for their shoulder in a primary care setting will be recruited to participate in a trial investigating the value of different exercise and education regimens. Patients that choose to participate will be randomized to 1 of 4 different treatment groups focused on strengthening of the rotator cuff and shoulder girdle muscles: eccentric strengthening alone; traditional strengthening alone; eccentric strengthening plus education focused on pain neuroscience, traditional strengthening plus education focused on pain neuroscience. All patients will be seen in the clinic for 4-6 sessions over a 4-week period, as well receive a home exercise program that aligns with the exercise group there were randomized to.

One-year outcomes will be compared across all 4 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65
2. Read and speak English well enough to provide informed consent, follow study instructions, and independently answer the questionnaires/surveys
3. TRICARE beneficiary (eligible for medical benefits in the Military Health System)
4. Primary complaint of new episode of unilateral shoulder pain; defined as not having sought care for shoulder condition in 6 months prior
5. Meets criteria for SAPS, as determined upon physical exam
6. At least 20% on either pain or disability subscales of the SPADI outcome measure
7. Available and willing to come in for treatment up to 8 sessions over a 4-week period

Exclusion Criteria:

1. History of shoulder dislocation, subluxation, fracture, adhesive capsulitis of the glenohumeral joint, or cervical/shoulder/upper back surgery, or shoulder injury as the result of trauma (e.g. fall, MVA)
2. Presence of cervical radiculopathy, radiculitis, or referral from cervical spine (reproduces shoulder symptoms)
3. Patient reports their condition is "acceptable" on Patient Acceptable Symptom State (PASS) at baseline
4. Anyone pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury
5. Unable to give informed consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 1 year
  This is a 100-point, 13-item self-administered questionnaire. It is divided into two subscales: a five-item pain subscale and an eight-item disability subscale. It is responsive to change and accurately discriminates between patients who are improving or worsening and has been reported to have a high test-retest reliability and internal consistency. A recent systematic review that compared four common shoulder questionnaires determined the SPADI was strongly correlated with the Disabilities of the Arm and Hand (DASH), American Shoulder and Elbow Surgeons (ASES) questionnaires and suitable for clinical use. The systematic review identified a minimal detectable change of 18 and a minimally clinically important difference of between 8-13 points.

SECONDARY OUTCOMES:
Patient Acceptable Symptom Scale (PASS) | 1 year
  Often defined as "the highest level of symptoms beyond which patients consider themselves well." This outcome measure has been used in previous studies looking at the effects of cervical thoracic thrust manipulation on shoulder pain. The question that will be asked to assess this level is, "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" Individuals who respond "yes" will be categorized as a success; thus, anyone reporting "yes" at baseline will be excluded from participation in the study. Between group differences at four time points will be assessed as percentage of subjects who find their current state acceptable, or answering "yes."
Patient Reported Outcomes Measurement Information System 57-Item Profile (PROMIS-57) v2.0 | 1 year
  The PROMIS 57 efficiently assesses several outcomes important to patients including pain intensity and interference, sleep disturbance, anxiety, depression, fatigue, and social role participation using items developed with rigorous methodology and patient input. This is a 57-item questionnaire with 8 questions per domain.
Revised Neurophysiology of Pain Questionnaire (NPQ) | 6 weeks
  The revised NPQ is a 12-item questionnaire that assesses a patient's understanding about pain and how it is produced in the body. The 12-item version was derived from the original 19-item Moseley Pain Questionnaire, after the removal of 7 items that did not function properly, and was found to have good test-retest reliability.
Survey of Pain Attitudes-35 (SOPA-35); 5-item Harm Scale | 1 year
  The full SOPA-35 is a 35-item shortened questionnaire from the original SOPA-57. The SOPA-35 Harm Scale is a subset of 5 items from the SOPA-35. This subset measures a person's belief that pain indicates damage and that activity can cause harm.
Healthcare Utilization | 2 years
  Shoulder-related healthcare costs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DPT, DSc, Principal Investigator — Director, Primary Care Musculoskeletal Research Center, Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data must go through a Data Sharing Agreement Application submitted and approved through the Defense Health Agency
Time Frame: DHA usually approves Data Sharing Agreements for 1 year at a time.
Access Criteria: Requires a Data Sharing Agreement Application to be submitted through the US Defense Health Agency
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Dejaco B, Habets B, van Loon C, van Grinsven S, van Cingel R. Eccentric versus conventional exercise therapy in patients with rotator cuff tendinopathy: a randomized, single blinded, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):2051-2059. doi: 10.1007/s00167-016-4223-x. Epub 2016 Jun 28. PMID 27351548
- [Background] Blume C, Wang-Price S, Trudelle-Jackson E, Ortiz A. COMPARISON OF ECCENTRIC AND CONCENTRIC EXERCISE INTERVENTIONS IN ADULTS WITH SUBACROMIAL IMPINGEMENT SYNDROME. Int J Sports Phys Ther. 2015 Aug;10(4):441-55. PMID 26346332
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Hanratty CE, McVeigh JG, Kerr DP, Basford JR, Finch MB, Pendleton A, Sim J. The effectiveness of physiotherapy exercises in subacromial impingement syndrome: a systematic review and meta-analysis. Semin Arthritis Rheum. 2012 Dec;42(3):297-316. doi: 10.1016/j.semarthrit.2012.03.015. Epub 2012 May 18. PMID 22607807
- [Background] Hsiao MS, Cameron KL, Tucker CJ, Benigni M, Blaine TA, Owens BD. Shoulder impingement in the United States military. J Shoulder Elbow Surg. 2015 Sep;24(9):1486-92. doi: 10.1016/j.jse.2015.02.021. Epub 2015 Apr 10. PMID 25865088